CLINICAL TRIAL: NCT06461910
Title: The Efficacy and Safety of Anti-PD-1 Combined With Thymalfasin and SOX in Neoadjuvant Treatment of cStage III Gastric or Gastroesophageal Junction Adenocarcinoma: A Prospective, Open-label, Single-arm, Phase II Clinical Study
Brief Title: Efficacy and Safety of Anti-PD-1, Thymalfasin, and SOX in Neoadjuvant Treatment of cStage III Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zekuan Xu (Other)
Responsible Party: Sponsor-Investigator, Zekuan Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GATES
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Esophagogastric Junction Adenocarcinoma
Keywords: neoadjuvant; PD-1; Thymalfasin; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Thymalfasin; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Serplulimab Combined with Thymalfasin and SOX (Experimental)
  Interventions: Drug: Serplulimab; Drug: thymalfasin; Drug: Oxaliplatin; Drug: Tegafur

INTERVENTIONS:
Drug: Serplulimab — 200 mg, i.v., D1, Q3W
Drug: thymalfasin — 4.8mg,sc,biw
Drug: Oxaliplatin — 130 mg/m2, i.v., D1, Q3W
Drug: Tegafur — oral administration: body surface area < 1.25, 40 mg each time; body surface area ≥ 1.25 to < 1.5, 50 mg each time; body surface area ≥ 1.5, 60 mg each time, twice daily for each treatment cycle at D1-D14

SUMMARY:
This Phase II clinical study is a prospective, open-label, single-arm trial designed to evaluate the efficacy and safety of combining anti-PD-1 therapy (Serplulimab) with thymalfasin and the SOX chemotherapy regimen as a neoadjuvant treatment for patients with clinical stage III gastric or gastroesophageal junction(GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm phase II clinical study to assess the efficacy and safety of Serplulimab in combination with thymalfasin and SOX regimen for neoadjuvant therapy of locally advanced gastric cancer. It is planned to enroll 30 patients with HER2-negative gastric or gastroesophageal junction adenocarcinoma confirmed by histopathology and/or cytology who were clinically staged as stage III resectable G/GEJ carcinoma as assessed by endoscopic ultrasonography, CT/MRI and other imaging. The primary endpoint of the study was pathological complete response (pCR) rate. The secondary end points included major pathological response(MPR) rate, Tumor Regression Grade (TRG), Clinical downstaging rate (T and/or N downstaging), Objective Response Rate (ORR), Disease Control Rate (DCR), R0 resection rate, Disease-free Survival (DFS), Overall Survival (OS) and treatment-related adverse events (TRAEs).

ELIGIBILITY:
Inclusion Criteria:

* Age and Diagnosis:

Patients aged 18-75 years with gastric (G) or gastroesophageal junction (GEJ) adenocarcinoma, regardless of gender.

* Stage and Diagnosis Confirmation:

According to the 8th edition of AJCC staging for gastric cancer, patients must be assessed via abdominal CT as cStage III (cT3-4aN1-3M0).

Diagnosis must be confirmed by endoscopy and pathology as G/GEJ adenocarcinoma (HER-2 negative).

Only patients with Siewert type III and type II (who do not require combined thoracic surgery) GEJ cancer are eligible.

* Surgical Assessment:

Tumors must be deemed resectable with curative intent (R0 resection) as determined by a gastrointestinal surgeon and a radiologist.

Patients must agree to undergo radical surgery and be deemed operable by a surgeon.

* Previous Treatments:

Patients must not have received prior systemic treatment for the current disease, including surgery, anti-tumor chemotherapy, radiotherapy, or immunotherapy.

* Survival Expectancy:

Expected survival of at least 3 months.

* Measurable Disease:

Tumors must be measurable according to RECIST v1.1 criteria.

* Performance Status:

ECOG PS score of 0-1 within 7 days prior to the first dose.

* Cardiac Function:

Good cardiac function, suitable for curative surgery. Preoperative evaluation by a cardiologist is required if there are clinical indications of underlying ischemic, valvular, or other severe heart diseases.

* Organ Function:

Normal function of major organs, meeting the following laboratory criteria:

Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without granulocyte colony-stimulating factor for the past 14 days.

Platelet count ≥ 100 x 10^9/L without transfusion for the past 14 days. Hemoglobin > 9 g/dL without transfusion or erythropoietin use for the past 14 days.

Total bilirubin ≤ 1.5 x upper limit of normal (ULN); if > 1.5 x ULN, direct bilirubin must be ≤ ULN.

AST and ALT ≤ 2.5 x ULN. Serum creatinine ≤ 1.5 x ULN and creatinine clearance (using Cockcroft-Gault formula) ≥ 60 ml/min.

Normal coagulation function (INR or PT ≤ 1.5 x ULN). Normal thyroid function (TSH within normal range, or normal T3/FT3 and FT4 if baseline TSH is out of range).

Normal myocardial enzyme spectrum (clinical judgment for non-significant lab abnormalities is acceptable).

* Weight:

Body weight ≥ 40 kg or BMI > 18.5.

* Female Patients:

Must be post-menopausal (no menses for at least one year without other causes) or surgically sterilized (removal of ovaries and/or uterus).

Women of childbearing potential must have a negative pregnancy test within 7 days prior to the first dose.

Agree to use highly effective contraception (annual failure rate < 1%) or abstain from heterosexual intercourse from the time of informed consent until at least 120 days after the last dose of the study drug or 9 months after surgery.

* Male Patients:

Must agree to use contraception or abstain from heterosexual intercourse from the time of informed consent until at least 120 days after the last dose of the study drug or 9 months after surgery.

Regular abstinence (e.g., calendar, ovulation, basal body temperature, or post-ovulation methods) and withdrawal are not acceptable forms of contraception.

* Informed Consent:

Patients must read, understand, and sign the informed consent form.

Exclusion Criteria:

* Other Malignancies:

Patients with a history of other malignancies within the past 5 years or concurrent malignancies. Exceptions include cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ prostate cancer, in situ cervical cancer, in situ breast cancer, stage I lung cancer, and stage I colorectal cancer.

Transplant Patients:

Patients planning to undergo or having previously undergone organ or bone marrow transplantation.

Blood Transfusions and Bleeding:

Patients who have received a blood transfusion within 2 weeks before the first dose, have a history of bleeding, or experienced any severe bleeding events (grade 3 or higher per CTCAE 4.0) within 4 weeks before screening.

Coagulation Disorders:

Patients with coagulation abnormalities and bleeding tendencies (INR > 1.5 without anticoagulants). Patients on anticoagulants or vitamin K antagonists like warfarin, heparin, or similar drugs can participate if INR ≤ 1.5, small-dose warfarin (1 mg/day) or aspirin (≤ 100 mg/day) is allowed for preventive use.

Thromboembolic Events:

Patients with arterial/venous thromboembolic events within 6 months before screening, such as stroke (including transient ischemic attacks), deep vein thrombosis (excluding cases resolved post-chemotherapy), and pulmonary embolism.

Cardiac Conditions:

Patients with myocardial infarction, uncontrolled arrhythmias (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females, using the Fridericia formula) within 6 months before the first dose.

NYHA class III-IV heart failure or LVEF < 50% on echocardiogram.

Proteinuria:

Urinalysis indicating proteinuria ≥ ++ and 24-hour urine protein > 1.0 g.

Oral Drug Absorption Issues:

Factors affecting oral drug absorption (e.g., inability to swallow, chronic diarrhea, bowel obstruction).

Pleural or Peritoneal Effusion:

Clinically significant pleural or peritoneal effusion requiring intervention.

HIV Infection:

Patients with HIV infection.

Active Tuberculosis:

Patients with active tuberculosis.

Non-Healing Wounds or Fractures:

Patients with long-standing unhealed wounds or incomplete healing of fractures.

Lung Diseases:

Patients with interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severely impaired lung function that could interfere with the detection and treatment of suspected drug-related pulmonary toxicity.

Autoimmune Diseases:

Patients with known active or suspected autoimmune diseases, except those in a stable state without systemic immunosuppressive treatment.

Chronic Autoimmune Diseases:

Severe chronic autoimmune diseases such as systemic lupus erythematosus; patients with a history of ulcerative colitis, Crohn's disease, or irritable bowel syndrome; history of sarcoidosis or tuberculosis; active hepatitis B or C, and HIV infection.

Well-controlled non-severe autoimmune diseases like dermatitis, arthritis, psoriasis can be included. Patients with hepatitis B virus titers < 500 copies/ml can participate.

Immunosuppressive Treatment:

Patients requiring systemic corticosteroids (> 10 mg/day prednisone equivalent) or other immunosuppressive drugs within 14 days before the first dose or during the study. Localized topical or inhaled steroids or adrenal hormone replacement therapy (≤ 10 mg/day prednisone equivalent) are allowed.

Active Infections:

Active infections requiring systemic treatment within 14 days before the first dose. Preventive antibiotic treatment (e.g., for urinary tract infection or COPD) is allowed.

Live Vaccines:

Patients who have received live vaccines within 28 days before the first dose. Inactivated viral vaccines for seasonal flu are allowed.

Previous Checkpoint Inhibitors:

Patients previously treated with checkpoint inhibitors like PD-1, PD-L1, or CTLA-4 inhibitors.

Immunomodulatory Treatments:

Patients who received immunomodulatory treatments (e.g., thymopentin, thymalfasin, interferons, CAR-T therapy) within 6 months before the first dose.

Other Clinical Studies:

Patients currently receiving other clinical study treatments or planning to start this study treatment within one month of completing a previous clinical study treatment.

Drug Allergies:

Known allergy or intolerance to any study drug or its components.

Substance Abuse:

History of alcohol, drug, or substance abuse. Patients who have stopped drinking can be included.

Compliance Issues:

Patients who are non-compliant with medical instructions, prescribed medications, or have incomplete records affecting efficacy or safety assessments.

Pregnancy and Breastfeeding:

Pregnant or breastfeeding women.

High-Risk Factors:

Patients with conditions increasing the risk of study participation or study drug use, or other severe, acute, or chronic diseases deemed unsuitable by the investigator.

Investigator Discretion:

Any other conditions that the investigator deems unsuitable for the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
pathological Complete Response (pCR) | from preoperative to 10 days postoperative
  pCR was defined as no residual tumor cells on the histologic examination of surgical specimens.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | from preoperative to 10 days postoperative
  For patients with surgically resectable gastric cancer after neoadjuvant therapy, the proportion of patients with less than 10% residual tumor cells in the primary site.
Tumor Regression Grade (TRG) | from preoperative to 10 days postoperative
  It is intended to grade the pathological response of tumor after neoadjuvant therapy and generally divide the grade mainly according to the proportion of fibrosis and residual tumor in the tumor. In this study, Becker criteria are used to grade TGR as follows: TRG1a (no residual tumor), equivalent to pCR; TRG1b (< 10% residual tumor); TRG2 (10% to 50% residual tumor); and TRG3 (> 50% residual tumor).
Clinical downstaging rate (T and/or N downstaging) | before surgery
  ypT0 ratio, ypN0 ratio, and preoperative imaging clinical stage will be counted, respectively, to compare with baseline imaging clinical stage downstaging ratio
Objective Response Rate (ORR) | before surgery
  It refers to the proportion of patients whose tumor shrinks to a certain extent and remains for a certain period of time, including CR (Complete Response) and PR (Partial Response) cases. Objective tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria).
Disease Control Rate (DCR) | before surgery
  It refers to the percentage of confirmed complete response (CR), partial response (PR) and stable disease (SD) cases among evaluable efficacy patients.
Disease-free Survival (DFS) | 2 years after surgery
  Disease-free survival refers to the time from the start of randomization to disease recurrence or death due to disease progression. DFS will be defined as the last date the patient is last confirmed to be disease-free survival if the patient does not experience disease progression during the study.
Overall Survival (OS) | 2 years after surgery
  Overall survival refers to the date from enrollment to death due to any cause.
R0 resection rate | from preoperative to 10 days postoperative
  R0 resection rate refers to the proportion of patients who complete R0 resection in surgically resectable patients after neoadjuvant therapy.
treatment-related adverse event (TRAE) | from the start of neoadjuvant therapy to 30 days after surgery
  incidence of treatment-related adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws.